CLINICAL TRIAL: NCT00679718
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled, Dose-Ranging Study of Multiple Ocular Instillations of INS365 Ophthalmic Solution vs. Placebo in Patients With Moderate to Severe Dry Eye Disease
Brief Title: A Study of INS365 Ophthalmic Solution in Patients With Moderate to Severe Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-103
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — diquafosol; Ophthalmic Solutions

INTERVENTIONS:
Drug: diquafosol tetrasodium (INS365) ophthalmic solution

SUMMARY:
To evaluate the efficacy and safety of INS365 Ophthalmic Solution when applied topically in patients with moderate to severe dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity of at least +0.7 ETDRS
* Six month history of dry eye disease
* Mild severity in two out of five symptoms
* Unanesthetized Schirmer score of less than or equal to 7mm
* Corneal fluorescein staining greater than or equal to 4 out of 15 or lissamine green conjunctival staining of greater than or equal to 5 out of 18

Exclusion Criteria:

* Nasal stimulated Schirmer score of less than 3mm
* Have ongoing ocular infection
* Have congenitally absent meibomian or lacrimal glands
* Have had punctal occlusion within a specified time prior to study
* Wear contact lens and refuse to remove them
* Have other excluded eye conditions.

Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2000-01; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Schirmer scores
Corneal staining
Conjunctival staining
Tear break-up time
Change in artificial tear usage
Patient-reported improvement of foreign body sensation

SECONDARY OUTCOMES:
Visual acuity
Investigator global severity assessment
Patient-reported dry eye symptoms other than foreign body sensation
Biomicroscopy
Ophthalmoscopy
IOP

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director, Study Director — Merck Sharp & Dohme LLC